CLINICAL TRIAL: NCT03071718
Title: Diet-induced Arrangement of the Gut Microbiome for Improvement of Cardiometabolic Health
Acronym: DINAMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paola Vitaglione (Other)
Responsible Party: Sponsor-Investigator, Paola Vitaglione, Associate Professor, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Federico II University
Record Dates: First submitted 2017-02-22; First posted 2017-03-07 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Overweight; Obesity
Keywords: cardiovascular diseases; gut microbiota; Mediterranean diet
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Med-D (Experimental): Subjects will follow a Mediterranean diet for two months
  Interventions: Other: Mediterranean diet
- Cont-D (Active Comparator): Subjects will follow a control diet for two months
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Mediterranean diet — Subjects in the Med-D group will be assigned a personalized diet prepared on the basis of own eating habits as established by 7-d food diary recalls. Energy values of habitual diets will be kept unchanged during Med-D intervention. Briefly, Med-D will be prepared so as to achieve a weekly consumption of:
  * 7 portions of milk or yogurt plus whole grain cereals,
  * 7 portions of nuts (30g)
  * At least 3 portion of absolute legumes
  * 14 portions of vegetables
  * 21 portions of fruit
  * 4 portions of whole grain pasta
  * 3 portions of whole grain pasta with vegetables or legumes
  * 7 portions of whole grain bread
  * 3 portions of fish
  * Extravirgin olive oil as unique source of discretional fats All subjects will be requested not to change physical activity levels during the 8 week intervention period.
  Arms: Med-D
Other: Control Diet — Control subjects will not change their habitual diet during intervention. All subjects will be requested not to change physical activity levels during the 8 week intervention period.
  Arms: Cont-D

SUMMARY:
Mediterranean diet (Med-D) has been recognized as an intangible cultural heritage by UNESCO and was shown to be beneficial for the treatment of obesity, type-2 diabetes and cardiovascular diseases. Individuals with the highest adherence to Med-D (classified according to Sofi et al., 2010) were characterized by increased levels of specific fibre-degrading bacteria, increased faecal levels of short chain fatty acids, and lower urinary concentrations of the atherogenic compound TMAO. However, the interplays between Med-D and microbial populations in the intestine remain unclear. Moreover, a number of clinical conditions like obesity, T2D, and atherosclerosis are associated with dysbiotic microbial ecosystems in the gut, i.e., shifts in the structure and function of the microbiota, but the characteristic features of dysbiotic gut communities and the impact of diet are not very well defined. The present study will evaluate the impact of Med-D on cardiometabolic health in human subjects via modification of intestinal microbial communities and its impact on health outcomes, mainly related to inflammatory, oxidative and hormonal status, in overweight subjects.

DETAILED DESCRIPTION:
It is estimated that in 2050 approximately 40-50% of the adult population worldwide will be overweight/obese (BMI > 25/30 kg/m2), with 10-20% of them developing insulin resistance resulting in metabolic syndrome and type-2 diabetes (T2D). T2D is forecast to become the 7th leading cause of death worldwide by 2030. Obesity and T2D are major risk factors for the development of cardiovascular diseases CVD. Despite currently available therapeutic strategies to reduce cardiovascular risk, less than one third of all cardiovascular events can be prevented. Hence, cardiovascular complications associated with obesity and metabolic syndrome/T2D are major health issues in Western societies, representing a substantial societal and economic burden (40 % of all deaths in Europe and EUR 196bn/y) that cannot be solved by the currently available treatment paradigms. Based on the close relation between CVD and diabetes mellitus, these two diseases together are referred to as cardiometabolic diseases (CMD). With respect to prevention strategies, it is crucial to understand molecular mechanisms that regulate transition phases from obesity and T2D to CVD. In particular, environmental factors (primarily diet and gut microorganisms) that promote or retard the development of cardiovascular complications must be identified in order to propose novel preventive strategies for maintaining cardiovascular health. Recent data showed that the communities of microorganisms in the intestine (gut microbiota) have a substantial impact on systemic cardiometabolic regulation, inflammatory activation and eventually CVD. Defining diet-microbiome profiles that contribute to resistance towards CMD development would be a major step forward in the field of nutritional disease prevention. Western dietary patterns, characterized by high consumption of red and processed meat, refined cereals and sugars, and high-fat dairy products, have been associated with a high incidence of CMD in Western countries. In contrast, the Mediterranean diet (Med-D) is a nutritionally recommended dietary pattern characterized by high-level intake of fruit, vegetables, legumes, nuts, minimally processed cereals, moderately high consumption of fish, low intake of saturated fat, meat and dairy products, regular but moderate consumption of alcohol and extra virgin olive oil as the main fat. Med-D has been recognized as an intangible cultural heritage by UNESCO (www.unesco.org/culture/ich/RL/00884) and was shown to be beneficial for the treatment of obesity, T2D, and CVD. Moreover, data from an Italian observational study including 153 subjects with different dietary regimens (omnivores, vegetarians, vegans) showed that individuals with the highest adherence to Med-D (classified according to Sofi et al., 2010) were characterized by increased levels of specific fibre-degrading bacteria, increased faecal levels of short chain fatty acids, and lower urinary concentrations of the atherogenic compound TMAO. However, the interplays between Med-D and microbial populations in the intestine remain unclear.

In this framework, the present project will focuses on the impact of diet on maintaining cardiometabolic health in human subjects via modification of intestinal microbial communities. Specific aims of the study are to establish new targeted intervention for maintenance of cardiometabolic health and thereby test the causal relationship between diet and the gut microbiome; to study the functionality of the intestinal milieu via meta-omics approaches, aiming at harmonization via standardization effort. The study will includes the establishment of a 2-months dietary intervention with an isocaloric Mediterranean diet (Med-D). Coupled with detailed host phenotyping and gut microbiota profiling during and after intervention, this will allow assessment of the causal effects of diet and the gut microbiome in populations at high risk for CVD.

Subjects in the Med-D group will be assigned a personalized diet prepared on the basis of own eating habits as established by 7-d food diary recalls. Energy values and whole macronutrient composition of habitual diets will be kept unchanged during Med-D intervention. However, changes in carbohydrate (dietary fibre vs. starch), dietary fat (saturated vs. mono/polyunsaturated fatty acids), and protein (vegetable vs. animal) composition will be applied. Briefly, Med-D will be prepared so as to achieve: 1) 2 % increase in energy from dietary fibre, mainly by replacing refined wheat products with wholegrain wheat products and/or with fruit/vegetables; 2) a repartition of energy from fat 1:3:1 (saturated : monounsaturated : polyunsaturated), replacing animal by vegetable fat and introducing/increasing virgin olive oil consumption; 3) a repartition of energy from proteins 1:4 (animal : vegetable proteins), replacing meat and/or dairy products by legumes. Control subjects will not change their habitual diet during intervention. All subjects will be requested not to change physical activity levels during the 8 week intervention period. Compliance will be assessed every 2 weeks by self-recorded 4-d (3 working and 1 weekend days) food diaries and by International Physical Activity Questionnaire (IPAQ). At baseline, after 1 month and after 2 months from starting the protocol, blood drawings will be performed and urine and feces will be collected from fasting subjects.

In a subgroup of participants the postprandial blood glucose and lipid response will be evaluated after a test meal resembling the lunch of the Mediterranean or the Control diet according to the assigned diet. Test meals will be performed at baseline and at the end of the intervention with samples taken at fasting and for 4 hours after the meal for determination of glucose, insulin, lipids, and SCFA.

Further analysis of compliance will be conducted based on metabolomics, allowing discrimination of animal/vegetable protein, olive oil intake and increased intake of foods with phenolics. Metabolomes (well known to reflect both diet and microbial metabolism) will also be compared between categories in order to identify protective or risk profiles using both bioinformatics and chemometrics approaches. Metagenomes will be analysed following SOPs utilized in landmark studies already published. Comparison of pre-defined groups of individuals will allow identification of microbial genes that have different abundances in the groups (e.g. twins discordant for CMD). Further, genes will be associated to continuous variables of clinical and nutritional interest (e.g. insulin sensitivity, intake of specific dietary components) by covariance analysis. Concatenated datasets of physiological output data, metagenomic and metabolome profiles from the intervention studies to predict subsets of features by multivariate analysis (PLS-DA) that can classify subjects according to their relative adherence to a Med-D. The profile will be used to probe the microbiome for specific alterations as a function of the interventions.

The sample size needed to detect an effect of Med-D on individual antioxidant and inflammatory markers is defined on the basis of a previous study conducted by UNINA showing that 30 participants in each treatment group would give sufficient power (a-error 0.05, 80% power, 2-sided testing) to detect a 50% change in urinary and fecal ferulic acid and a 30% change of fasting TNF. In addition, it is estimated that a sample size of 28 participants would be adequate to detect a 10% change in fasting total cholesterol by using variation in accordance with other studies. The number of participants will be increased to 40 per group to compensate for dropouts. Samples (faeces, venous blood, and non-acidified 24h urine) will be collected at baseline, 4 and 8 weeks after starting dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

Subject will be selected by interviews on health status, dietary and behavioural lifestyle factors, anthropometric data and a 7-d food diary recall.

Inclusion criteria are:

* men and women aged 18-65;
* BMI>24kg/m2;
* a diet characterized by low adherence to Med-D, with absence of any food supplements and alternative medication;
* intake of fruit/vegetables < 3 servings/d;
* a low level of physical activity (< 500 metabolic equivalent min/week).

Exclusion Criteria:

* Subjects having any chronic or metabolic diseases, food allergies, or following a dietary regimen or medication <3 months preceding the study will be excluded.
* Participation in other clinical trials, pregnancy or lactation are also exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Changes in fasting plasma lipids | 2months
  Measure of plasma concentrations (mg/dL) of Total-, LDL-, and HDL-Cholesterol, as well as Triglycerides
Changes in faecal levels of short chain fatty acids | 2months
  measure of short chain fatty acids from faecal samples

SECONDARY OUTCOMES:
Changes in faecal microbiome | 2months
  Measure of faecal microbiome
Changes in urinary TMAO concentration | 2months
  measure of urinary TMAO (μM)
Variation of serum polyphenols concentration | 2months
  Measure of serum polyphenols concentration (nmol/L)
Variation of serum gastro-intestinal hormone concentration | 2months
  Measure of plasma GLP-1 concentrations (mg/dL)
Variation of serum gastro-intestinal hormone concentration | 2months
  Measure of plasma GIP concentrations (mg/dL)
Variation of serum gastro-intestinal hormone concentration | 2months
  Measure of plasma Glucagon concentrations (mg/dL)
Variation of serum gastro-intestinal hormone concentration | 2months
  Measure of plasma Ghrelin concentrations (mg/dL)
Variation of serum gastro-intestinal hormone concentration | 2months
  Measure of plasma Insulin concentrations (mg/dL)
Variation of plasma endocannabinoids concentration | 2months
  Measure of plasma endocannabinoids concentrations (mg/dL)
Variation of blood pressure | 2months
  Measure of blood pressure (mmHg)
Changes in fasting inflammatory blood markers | 2months
  Measure of plasma C-reactive protein (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vitaglione, Professor, Study Director — Department of Agricultural Sciences, Federico II University; Danilo Ercolini, Professor, Study Chair — Department of Agricultural Sciences, Federico II University; Angela Rivellese, Professor, Principal Investigator — Department of Clinical and Experimental Medicine, Federico II University; Ilario Mennella, PhD, Principal Investigator — Department of Agricultural Sciences, Federico II University
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We will decide as soon as we will have data analysis completed and a clear idea on publication rute according with the other coauthors.

REFERENCES:
- [Derived] Tagliamonte S, Laiola M, Ferracane R, Vitale M, Gallo MA, Meslier V, Pons N, Ercolini D, Vitaglione P. Mediterranean diet consumption affects the endocannabinoid system in overweight and obese subjects: possible links with gut microbiome, insulin resistance and inflammation. Eur J Nutr. 2021 Oct;60(7):3703-3716. doi: 10.1007/s00394-021-02538-8. Epub 2021 Mar 24. PMID 33763720

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03071718/Prot_SAP_000.pdf